CLINICAL TRIAL: NCT00197353
Title: Sympathectomy-Mediated Vasodilatation and Differential Sensory Block After Epidural Bupivacaine: a Randomized Concentration Ranging Study
Brief Title: Study of Different Concentrations of Epidural Bupivacaine for the Effects on Vasodilatation and Sensory Block
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PPG1-ginosar-HMO-CTIL
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2005-05

CONDITIONS: Intraoperative Complications
Keywords: Anesthesia, Epidural; Pharmacology; Dose-Response Relationship, Drug; Sympathectomy; Photoplethysmography
MeSH Terms: conditions — Intraoperative Complications

INTERVENTIONS:
Drug: Epidural bupivacaine (dose/concentration/volume ranging)

SUMMARY:
This study aims to compare human subjects receiving epidural bupivacaine local anesthetic at different doses and concentrations and to assess the effect on vasodilatation (sympathectomy), sensory and motor block.

The hypothesis is that the drug concentration is more important than drug dose in the determination of the extent and intensity of differential sympathetic, sensory and motor block following epidural local anesthetic.

DETAILED DESCRIPTION:
There is controversy regarding the factors that determine the extent and intensity of epidural drug action. Most studies have focused on the inter-related triad of dose, concentration and volume.

We compare three groups: group A: 10ml of 0.5% bupivacaine; group B: 10ml of 0.25% bupivacaine and group C: 40ml of 0.0625% bupivacaine. When comparing these groups, groups A & B have the same volume of epidural drug, and groups B & C have the same total dose.

In particular this study compares different methods of assessing the sympathetic block (causing vasodilatation). These methods include skin temperature changes, hemodynamic changes and photoplethysmography.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for extracorporeal shock wave lithotripsy (ESWL) under epidural anesthesia between March to September 1999

Exclusion Criteria:

* graded as ASA 3 or higher, below 18 or above 70 years of age, if they had peripheral vascular disease, baseline neurological deficit, or had any other contraindication for regional anesthesia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 1999-03; Study Completion 1999-09

PRIMARY OUTCOMES:
Index of sympathectomy: photoplethysmography derived amplitude-baseline ratio from foot and hand; data measured at time 0, 5, 10 and 20 min following epidural; data expressed as % change from baseline and as area under time effect curve.

SECONDARY OUTCOMES:
1. Other indices of sympathectomy:
a. Photoplethysmography derived baseline change (ln (Blepi/Blo));
b. Photoplethysmography derived time lag between pulse reaching hand and foot;
c. Blood pressure (mean, systolic, diastolic);
d. Skin temperature changes (finger and toe temperature change from baseline, toe-thigh and finger-arm temperature gradients).
2. Sensory level (pinprick, touch, cold)
3. Motor block (Bromage scale)
All assessments made at 0, 5, 10 and 20 minutes after epidural drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Ginosar, BSc MBBS, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Hebrew University Medical Center, Jerusalem, Israel

REFERENCES:
- [Result] Babchenko A, Davidson E, Ginosar Y, Kurz V, Faib I, Adler D, Nitzan M. Photoplethysmographic measurement of changes in total and pulsatile tissue blood volume, following sympathetic blockade. Physiol Meas. 2001 May;22(2):389-96. doi: 10.1088/0967-3334/22/2/310. PMID 11411248
- [Derived] Ginosar Y, Weiniger CF, Meroz Y, Kurz V, Bdolah-Abram T, Babchenko A, Nitzan M, Davidson EM. Pulse oximeter perfusion index as an early indicator of sympathectomy after epidural anesthesia. Acta Anaesthesiol Scand. 2009 Sep;53(8):1018-26. doi: 10.1111/j.1399-6576.2009.01968.x. Epub 2009 Apr 24. PMID 19397502
- [Derived] Ginosar Y, Weiniger CF, Kurz V, Babchenko A, Nitzan M, Davidson E. Sympathectomy-mediated vasodilatation: a randomized concentration ranging study of epidural bupivacaine. Can J Anaesth. 2009 Mar;56(3):213-21. doi: 10.1007/s12630-008-9036-z. Epub 2009 Jan 28. PMID 19247742